CLINICAL TRIAL: NCT05927324
Title: Can Clinician Assisted Videofeedback Exposure Approach Therapy (CAVEAT) Help Post-traumatically Stressed Mothers Change Their Mind About Their Toddlers?
Brief Title: Clinician-Assisted Videofeedback Exposure-Approach Therapy (CAVEAT) Trial
Acronym: CAVEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: International Psychoanalytical Association (Unknown)
Responsible Party: Principal Investigator, Daniel Schechter, Associate Professor of Psychiatry, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPECTRE-CAVEAT
Record Dates: First submitted 2023-05-30; First posted 2023-07-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Interpersonal Violence; PTSD; Women; Infants and Children; Attachment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental): CAVEAT active treatment group
  Interventions: Behavioral: CAVEAT

INTERVENTIONS:
Behavioral: CAVEAT — Brief psychotherapy with mothers of infants and young children, to which infants and young children attend many but not all sessions with mother

SUMMARY:
The first study proposed is a small (n= 10 to 12 maximum) open feasibility trial of CAVEAT which is a 16-session manualized brief psychotherapy prototcol that is designed to help mothers of infants and young children, whereby the mothers have been exposed to interpersonal violence (i.e. childhood maltreatment and family violence, intimate and non-intimate partner violence, interpersonal combat and or other forms of terrorism or political violence including physical and sexual assault) and who have developed related post-traumatic stress. The treatment uses an integration and extension of evidence-based techniques: Modified Interaction Guidance, Prolonged Exposure Therapy for PTSD, Child-Parent Psychotherapy, and Minding the Baby, in order to help mothers with post-traumatic dysregulation and difficulty in their maintaining sensitivity during challenging parent-child interactions (i.e. when mothers are confronted with child helpless states, emotion dysregulation, negative affect and child aggression). Outcome measures will initially include: maternal attributions towards her child (i.e. perception of child's personality), maternal-child behavior, and maternal-child symptoms of attachment disturbance and PTSD. This feasibility study is meant to perfect the manual and to prepare for an initial open trial with a larger clinical sample including analysis of pre- and post-intervention measures before further randomized control study can be done.

DETAILED DESCRIPTION:
1. SYNOPSIS OF THE STUDY Sponsor / Sponsor-Investigator Sponsor: Prof. Kerstin von Plessen Sponsor-Investigator: Prof. Daniel S. Schechter Investigator: Mrs. Sandra Rusconi Serpa, MSc, FSP Study Title Feasibility of a brief manualized psychotherapy for traumatized mothers and their young children: Clinician Assisted Videofeedback Exposure Approach Therapy (CAVEAT) Short Title / Study ID CAVEAT Feasibility Study Protocol Version and Date Version 1.0, DATE Study registration Registered on international register (clinicaltrial.gov) provisionally Study category and Rationale This feasibility study conforms to a clinical trial of category A Background and Rationale The present study aims to determine if the manualized brief psychotherapy "Clinician Assisted Videofeedback Exposure-Approach Therapy (CAVEAT)" can be administered to violence-exposed mothers and their young children (ages 1-5 years) in the ambulatory care center of a Swiss public hospital (SUPEA, CHUV) during a psychotherapy of 16 sessions. CAVEAT is based on an amalgam of four existing evidence-based psychotherapy models (Child-Parent psychotherapy, Parental Mentalization, Interaction Guidance, Prolonged Exposure) for parents, infants and young children and traumatized adults that led to the novel, core therapeutic technique developed by Prof. Schechter and colleagues "Clinician Assisted Videofeedback Exposure Session(s) or "CAVES" which has been shown to be successful in positively altering mothers' perception of their young children in two open trials. From the existing literature, the investigataors know that parent-child relationship-based psychotherapies improve significantly maternal sensitivity to their child's communication, which is in part based on maternal capacity to perceive more accurately the young child's emotional communication and to take the child's perspective. Moreover, dyadic psychotherapy models using video-feedback and support of parental mentalization have been shown across models more generally to improve the quality of mother-child interaction.

Risk / Benefit Assessment The risks of participating in this study are estimated as minimal (category A). The proposed intervention involves standard, validated psychotherapeutic procedures with the addition of clinician-assisted videofeedback exposure to naturalistic challenges that are typically stressful for young children and that are "in situation" by the clinician in collaboration with the child's mother during the filmed parent-child interaction sessions. This latter technique has been used without complication in both mental health referred and non-referred pediatrics samples with positive clinical effects in both studies. The investigators estimate that the risks of such an intervention are therefore limited. Though, if a matter arises that is severe, urgent or cannot be dealt with in the psychotherapy as conceived in the model, based on the therapist assessment, proper interventions and/or referrals will be made. Regarding the potential benefits

1. An increase in maternal ability to take her very young child's perspective
2. To respond more sensitively to the child's developmental needs and emotional communication,
3. To be aware of what triggers post-traumatic stress during parent-child interactions,
4. Reduction in re-experiencing, avoidance, negative cognitions, and hyperarousal in day-to-day life with one's child
5. Acquisition of increased tools for self and mutual regulation and stress-reduction during are benefits of participating in the study.

If this form of manualized psychotherapy proves feasible to administer in a public hospital outpatient mental health clinic for children, it could potentially be implemented for this group of patients in a study that tests its efficacy in terms of improvement in parental stress, maternal sensitivity, and reduction of parent-child relational disturbance, potentially benefitting the larger group of these difficult-to-treat child-parent dyads.

Objective(s) The aim of the submitted study is to determine whether the manualized, brief child-parent psychotherapy CAVEAT can be feasibly performed in a child and adolescent psychiatric ambulatory care center at the CHUV, a public university-hospital, this with child and mothers who have experienced IPV and who present to the clinic with concerns about their child's risk for emotional and/or behavior difficulties and/or who note relational disturbances with their very young children ages 1-5 years and/or problems with their parenting.

Aim 1: To assess the feasibility of the recruitment procedures and adherence to treatment among patients, mother, and child therapeutic alliance as well as in terms of the mother and child satisfaction.

Aim 2: To assess if CAVEAT evaluation measures (questionnaires and observed interactions) will be found appropriate, adequate, and sensitive by patients and therapists to the outcomes targeted Aim 3: To assess if CAVEAT for the therapists is feasible to administer in terms of the application of the psychotherapy manual and the psychotherapy procedures involved to the clinic population.

Study Design Open-trial feasibility study. Interim, and post-treatment measures of patient and therapist satisfaction and patient-therapist therapeutic alliance and agreement on treatment goals and realization of treatment objectives. Counts of number of completed sessions and drop-outs before completing the full course of therapy will be noted as well as the clinical supervisor's assessment of therapist adherence to the CAVEAT manual.

Statistical Considerations As this is an open feasibility study of 12 participant-dyads only, results will be in terms of descriptive statistics, counts, and percentages.

Control Intervention: There is no control group or intervention in this pilot feasibility study.

Study procedures As a feasibility study, the present study will implement and check the procedures related to recruitment; inclusion, retention vs drop-out; questionnaire completion and interviews; recording and transcription.

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers of infants and young children ages 12-54 months
* Mothers and infants have lived together most of the child's life from the time of birth

Exclusion Criteria:

* Actively psychotic or substance-abusing mothers;
* Mothers and/or children who are physically or mentally handicapped so as to prevent adequate participation in required research tasks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire | through study completion, an average of 1 year
  Parental and Therapist individual self-report questionnaire

SECONDARY OUTCOMES:
Parenting Stress Questionnaire-Short Form | through study completion, an average of 1 year
  Parental self-report questionnaire
Maternal Attributions Rating Scale | through study completion, an average of 1 year
  Clinician rating of parental attributions towards the child with scores ranging from 10-50, higher scores representing worse outcome (more negative and age-inappropriate attribution by clinician rating)

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Yes

REFERENCES:
- [Background] Schechter DS, Moser DA, Reliford A, McCaw JE, Coates SW, Turner JB, Serpa SR, Willheim E. Negative and distorted attributions towards child, self, and primary attachment figure among posttraumatically stressed mothers: what changes with Clinician Assisted Videofeedback Exposure Sessions (CAVES). Child Psychiatry Hum Dev. 2015 Feb;46(1):10-20. doi: 10.1007/s10578-014-0447-5. PMID 24553738
- [Background] Schechter DS, Myers MM, Brunelli SA, Coates SW, Zeanah CH, Davies M, Grienenberger JF, Marshall RD, McCaw JE, Trabka KA, Liebowitz MR. Traumatized mothers can change their minds about their toddlers: Understanding how a novel use of videofeedback supports positive change of maternal attributions. Infant Ment Health J. 2006 Sep;27(5):429-447. doi: 10.1002/imhj.20101. PMID 18007960
- See also: Link to CAVEAT concept introduction article (in German) — https://serval.unil.ch/fr/notice/serval:BIB_E777AA5BB11D